CLINICAL TRIAL: NCT00773604
Title: Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) in Patients With Dystonia
Brief Title: Deep Brain Stimulation in Patients With Dystonia
Acronym: STN DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Private donor
Record Dates: First submitted 2008-10-07; First posted 2008-10-16 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Dystonia
Keywords: blepharospasm; Deep brain Stimulation; cervical dystonia; cranial dystonia; generalized dystonia; subthalamic nucleus; DBS
MeSH Terms: conditions — Dystonia; Blepharospasm; Torticollis | interventions — Deep Brain Stimulation; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): Deep Brain Stimulation
  Interventions: Device: Medtronic implantable deep brain stimulation (DBS) system

INTERVENTIONS:
Device: Medtronic implantable deep brain stimulation (DBS) system — surgical placement of deep brain stimulation system for treatment of dystonia

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of deep brain stimulation (DBS) of the subthalamic nucleus (STN)for primary dystonia.

DETAILED DESCRIPTION:
Dystonia is an uncommon brain disorder in which there is abnormal muscle tone producing twisting, writhing movements and abnormal postures. It is associated with abnormal electrical activity in two groups of nerve cells in the brain called the globus pallidus internus (GPi) and the subthalamic nucleus (STN). Deep brain stimulation (DBS) has been shown to be an effective treatment in patients with medically refractory dystonia and is currently approved for both the GPi and STN targets under a humanitarian device exemption (HDE) for use in segmental and generalized primary dystonia as well as focal cervical dystonia. GPi DBS appears to be effective for medication-refractory focal and segmental dystonia affecting the cranial and cervical regions in open-label series, but recently GPi stimulation has been associated with subtle motor disturbances in previously non-dystonic body regions (i.e., arms and legs) in this population of patients. DBS of the STN has also been reported to be effective for treating generalized and cervical dystonia in small open label trials. STN DBS for cranial and cervical regions may provide similar efficacy in the treatment of dystonia as GPi DBS, but without unwanted stimulation-induced motor effects. Objectives of this study are to evaluate the safety and efficacy of STN DBS for dystonia. Up to twenty-five patients will be screened, consented, and enrolled in this study. All patients will undergo bilateral STN DBS for dystonia. Participants will be evaluated pre- and postoperatively with standard dystonia rating scale Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS), and a patient questionnaire will be administered postoperatively to determine if patients are experiencing stimulation-induced motor adverse effects and will be logged for safety monitoring. This pilot study will provide preliminary open label efficacy outcomes for STN DBS in the treatment of primary dystonia and will help determine if this target should be compared to GPi DBS in a larger double-blind trial.

ELIGIBILITY:
Inclusion Criteria:

* Refractory primary dystonia diagnosed by a movement disorders neurologist
* Severe functional impairment despite optimal medical management, including failed botulinum toxin therapy
* Age 7-80 years (UCSF patients) and 18-80 (VA patients)

Exclusion Criteria:

* Patients considered at high risk for elective neurosurgery because of co-morbid conditions
* Brain MRI showing extensive brain atrophy or small vessel ischemic disease
* Pregnancy
* Inability to tolerate awake microelectrode-guided neurosurgery
* Inability to follow up with post-operative study visits
* Inability to speak or read English
* Patients with a score of 4.5 or lower on the BFMDRS movement scale
* Patients with Secondary dystonia

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ostrem, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco Veterans Administration Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with research collaborators.
Time Frame: De-identified data may be available after results have been published, indefinitely.
Access Criteria: Research collaborations accepted by study investigators

REFERENCES:
- [Derived] Ostrem JL, San Luciano M, Dodenhoff KA, Ziman N, Markun LC, Racine CA, de Hemptinne C, Volz MM, Heath SL, Starr PA. Subthalamic nucleus deep brain stimulation in isolated dystonia: A 3-year follow-up study. Neurology. 2017 Jan 3;88(1):25-35. doi: 10.1212/WNL.0000000000003451. Epub 2016 Nov 30. PMID 27903810

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Cohort: This was a single arm open label study of 9 patients who were treated with STN DBS for isolated dystonia
Period: Overall Study
Arm/Group | Open Label Cohort
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Cohort
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 48.95 [17 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: The Toronto Western Spasmodic Rating Scale (TWSTRS) Movement Scores Measured Before DBS Surgery (Baseline) and at 12 Months
Description: Total TWSTRS score range is 0-88, where higher score indicates worse symptoms. Values are calculated by baseline minus 12 month, where higher difference score of change between baseline and 12 months means better outcome (more improvement)
Time Frame: Baseline and 12 months
Population: Patients implanted and treated with DBS
Measure: Mean (Full Range); unit: TWSTRS total score change
Arm/Group | Open Label Cohort
Number analyzed (Participants) | 9
TWSTRS total score change | 33.5 [9.2 to 57.75]

ADVERSE EVENTS:
Groups:
- Treatment: DBS treatment patients
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=9)
Dyskinesia (Nervous system disorders) | 8
Depression, transient worsening (Psychiatric disorders) | 5
Weight gain (Metabolism and nutrition disorders) | 4
Anxiety, worsened (Psychiatric disorders) | 2
Dysarthria (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
Transient erythema around parietal incision site (Skin and subcutaneous tissue disorders) | 1
Subgaleal cerebral fluid collection around burr-hole cap (Surgical and medical procedures) | 1
Persistent pain at IPG site (Surgical and medical procedures) | 1
Shock-like sensations (Nervous system disorders) | 1
Migraine headaches, worsened (Nervous system disorders) | 1
Sensory deficit in hand, worsened (Nervous system disorders) | 1
Lower extremity paresthesias (Nervous system disorders) | 1
Blood pressure instability (Blood and lymphatic system disorders) | 1
Fall (Nervous system disorders) | 1
Knee dislocation (Musculoskeletal and connective tissue disorders) | 1
Knee injury (Musculoskeletal and connective tissue disorders) | 1
Hip pain, worsened (Musculoskeletal and connective tissue disorders) | 1
Fourth cranial nerve palsy, preexisting (Nervous system disorders) | 1
Handwriting difficulties (General disorders) | 1
Humming sounds in ear, worsened (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No